CLINICAL TRIAL: NCT02476344
Title: Classification and Characterization of Physical Strains During Sorting Series: Physiological Aspects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-15-2188-OF-CTIL
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): 40 subjects will undergo the experiment protocol, total 3 days, each consisting different training exercises.
  Interventions: Other: experiment protocol

INTERVENTIONS:
Other: experiment protocol — each subject will perform the following 3 days experiment protocol, consisting of army training exercises:
  1. sack carrying exercise.
  2. crawling exercise.
  3. combined exercise: sack carrying, crawling and sprints.
  heart rate, core temperature, lactic acid and CPK levels will be monitored continuously.

SUMMARY:
2 young candidates have tragically died during army pre-recruitment sorting series in 2006. As part of the classification and characterization of the physical aspects of the training, this experiment was requested.

We aim at determining the characteristics of physical strains in sorting series, by objective and subjective parameters and evaluating the difficulty levels and intensity of those strains.

DETAILED DESCRIPTION:
each subject will perform the following 3 days experiment protocol, consisting of army training exercises:

1. sack carrying exercise; the subjects will go up and down through a steep slope with sand sack on their back (path length is 200 meters,10 repetitions).

   the first day will also include recruitment and medical examination, in addition to the exercise.
2. crawling exercise; the subjects will crawl with knee's protectors back and forth (path length is 20 meters,15 repetitions).
3. combined exercise: sprints session (path length 600 meter, 3 repetitions),15 min break, sack carrying session (same protocol as first day), 45 min break and crawling session (same protocol as the second day).

during all exercises heart rate, core temperature, lactic acid and CPK levels will be monitored continuously.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-22 years.
* Healthy civilian volunteers.
* without skeleton-muscle illnesses.
* without Infectious disease 2 weeks prior to the experiment.

Exclusion Criteria:

* any physical condition.
* physician decition.

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch) | 3 experiment days
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).

SECONDARY OUTCOMES:
CPK measured from blood sample (3ml) in the lab | 3 experiment days
  CPK levels will be measured from blood sample (3ml) in the lab
lactic acid measured using lactat-meter (Lactate pro LT-1710) | 3 experiment days
  lactic acid levels from finger blood (5ul) using lactat-meter (Lactate pro LT-1710)
body core temperature monitored using telemetry pill | 3 experiment days
  core temperature will be monitored using telemetry pill

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel